CLINICAL TRIAL: NCT01696396
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Efficacy of AMG 181 in Subjects With Moderate to Severe Crohn's Disease
Brief Title: Abrilumab (AMG 181) in Adults With Moderate to Severe Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20110232; 2012-000529-31 (EudraCT Number)
Record Dates: First submitted 2012-09-27; First posted 2012-10-01 (Estimated); Results first posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-05

CONDITIONS: Crohn's Disease
Keywords: IBD, Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — abrilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo Q4W/Abrilumab 210 mg Q3M (Placebo Comparator): Participants received placebo by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks thereafter until week 24.
  During the open-label period, participants received abrilumab 210 mg once every 3 months (Q3M) for 108 weeks.
  Interventions: Drug: Abrilumab; Drug: Placebo
- Abrilumab 21 mg Q4W/Abrilumab 210 mg Q3M (Experimental): Participants received 21 mg abrilumab by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks (Q4W) thereafter until week 24.
  During the open-label period, participants received abrilumab 210 mg once every 3 months (Q3M) for 108 weeks.
  Interventions: Drug: Abrilumab
- Abrilumab 70 mg Q4W/Abrilumab 210 mg Q3M (Experimental): Participants received 70 mg abrilumab by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks thereafter until week 24.
  During the open-label period, participants received abrilumab 210 mg once every 3 months (Q3M) for 108 weeks.
  Interventions: Drug: Abrilumab
- Abrilumab 210 mg/Abrilumab 210 mg Q3M (Experimental): Participants received a single dose of 210 mg abrilumab by subcutaneous injection on day 1, followed by placebo at week 2, week 4, and every 4 weeks thereafter until week 24.
  During the open-label period, participants received abrilumab 210 mg once every 3 months (Q3M)for 108 weeks.
  Interventions: Drug: Abrilumab; Drug: Placebo

INTERVENTIONS:
Drug: Abrilumab — Administered by subcutaneous injection.
  Other Names: AMG 181
Drug: Placebo — Placebo matching to abrilumab administered by subcutaneous injection
  Arms: Abrilumab 210 mg/Abrilumab 210 mg Q3M; Placebo Q4W/Abrilumab 210 mg Q3M

SUMMARY:
The primary objective of this study is to evaluate the efficacy of abrilumab as measured by the proportion of participants achieving Crohn's Disease Activity Index (CDAI) remission (CDAI < 150) after treatment for 8 weeks.

DETAILED DESCRIPTION:
The study consisted of a 24-week double-blind treatment period, a 108-week open-label treatment period, and a 2-year safety follow-up period.

Participants who did not reach minimal improvement, or experienced disease worsening after initial response, had the option to receive open-label abrilumab 210 mg every 3 months (Q3M) beginning at double-blind period week 12 or after. Not reaching minimal improvement was defined as not having an improvement in CDAI score of ≥ 70 points from baseline on 2 consecutive visits (at or after week 8) at least 2 weeks apart. Disease worsening after week 8 (or week 12) response was defined as having an increase in CDAI score of ≥ 70 points from the week 8 (or week 12) CDAI score on 2 consecutive visits at least 2 weeks apart, and a CDAI score of > 150.

Participants were planned to be randomized in a 2:1:2:1 ratio to SC placebo or abrilumab at 21 mg, 70 mg (on day 1, week 2, week 4, and every 4 weeks thereafter until week 24), or 210 mg (on day 1 followed by placebo in weeks 2 and 4 and every 4 weeks thereafter until week 24), respectively. Due to a consistent discrepancy between the investigational product (IP) instruction manual (IPIM) description of vial positions and the actual vial positions in the IP package participants were initially randomized to 3 arms (placebo, 70 mg, and 210 mg) with a randomization ratio of 3:2:1. The study was temporarily paused while this issue was investigated. Once the discrepancy was corrected, Protocol Amendment 3 implemented, and affected participants completed their double-blind treatment period, the study resumed enrollment and randomization per protocol. Neither the randomization nor study blind was compromised and therefore the intent-to-treat principle was maintained.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ileal, ileo-colonic, or colonic Crohn's disease for a minimum of 6 months prior to baseline
* Moderately to severely active Crohn's disease defined by a CDAI score ≥ 220 and ≤ 450 at baseline
* Evidence of active inflammation within 12 weeks prior to baseline
* Demonstrated an inadequate response to, loss of response to, or intolerance to at least one of the following agents: Immunomodulators and/or anti-tumor necrosis factor (TNF) agents or to corticosteroids (non-US sites only).
* Neurological exam free of clinically significant, unexplained signs or symptoms during screening and no clinically significant change prior to randomization
* Subject has no known history of active tuberculosis and has a negative test for tuberculosis during screening

Exclusion Criteria:

* Short bowel syndrome
* Stricture with obstructive symptoms within 3 months
* Bowel surgery within 12 weeks prior baseline, or has planned bowel surgery within 24 weeks from baseline
* Ileostomy and/or colostomy
* Any gastric or intestinal pouch
* Evidence of an infected abscess
* Bowel perforation or evidence of non-inflammatory obstruction during the 6 months prior to baseline
* Stool positive for C. difficile toxin at screening
* Any uncontrolled or clinically significant systemic disease
* Known to have tested positive for hepatitis B virus surface antigen, hepatitis C virus antibody, or human immunodeficiency virus (HIV)
* Any underlying condition that predisposes subject to infections
* Subject has malignancy (other than resected cutaneous basal or cutaneous squamous cell carcinoma, or treated in situ cervical cancer considered cured) within 5 years of baseline
* Received an anti-TNF agent, cyclosporine, mycophenolate mofetil, sirolimus (rapamycin), thalidomide, tacrolimus, topical (rectal) aminosalicylic acid (eg, mesalamine) or topical (rectal) steroids, intravenous or intramuscular corticosteroids within protocol-specified time periods.
* Any prior exposure to antagonists of integrins or integrin ligands (eg, natalizumab, efalizumab, or vedolizumab), rituximab, or TNF kinoid immunotherapies, AMG 181, or any form of cell-based transplantation
* Received treatment of infection with intravenous (within 30 days of baseline) or oral (within 14 days prior to baseline) antibiotics, antivirals, or antifungals
* Significant laboratory abnormalities
* Pregnant or breast feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2012-12-04 (Actual); Primary Completion 2014-12-26 (Actual); Study Completion 2018-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (78):
- United States (24):
  - Research Site, Birmingham, Alabama
  - Research Site, Dothan, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Goodyear, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, La Jolla, California
  - Research Site, Jacksonville, Florida
  - Research Site, Sanford, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Arlington Heights, Illinois
  - Research Site, Ann Arbor, Michigan
  - Research Site, Chesterfield, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Mexico, Missouri
  - Research Site, Great Neck, New York
  - Hospital, New York, New York
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Mentor, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Germantown, Tennessee
  - Research Site, Seattle, Washington
- Austria (3):
  - Research Site, Innsbruck
  - Research Site, Sankt Veit an der Glan
  - Research Site, Vienna
- Belgium (4):
  - Research Site, Bonheiden
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Leuven
- Canada (7):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Greater Sudbury, Ontario
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Saskatoon, Saskatchewan
- Czechia (3):
  - Research Site, Hradec Králové
  - Research Site, Prague
  - Research Site, Ústí nad Labem
- Denmark (6):
  - Research Site, Aalborg
  - Research Site, Århus C
  - Research Site, Herlev
  - Research Site, Hvidovre
  - Research Site, Køge
  - Research Site, Odense C
- France (8):
  - Research Site, Amiens
  - Research Site, Caen
  - Research Site, Clichy
  - Research Site, Lille
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Vandœuvre-lès-Nancy
- Germany (4):
  - Research Site, Hamburg
  - Research Site, Leipzig
  - Research Site, Minden
  - Research Site, Stuttgart
- Hungary (5):
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Miskolc
  - Research Site, Szekszárd
- Netherlands (5):
  - Research Site, Amsterdam
  - Research Site, Breda
  - Research Site, Leiden
  - Research Site, Maastricht
  - Research Site, Rotterdam
- Switzerland (3):
  - Research Site, Basel
  - Research Site, Bern
  - Research Site, Zurich
- United Kingdom (6):
  - Research Site, Birmingham
  - Research Site, Coventry
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Norwich
  - Research Site, Torquay

REFERENCES:
- [Background] Dummer R, Hoeller C, Gruter IP, Michielin O. Combining talimogene laherparepvec with immunotherapies in melanoma and other solid tumors. Cancer Immunol Immunother. 2017 Jun;66(6):683-695. doi: 10.1007/s00262-017-1967-1. Epub 2017 Feb 25. PMID 28238174
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 84 centers in Canada, European Union, and the United States. Participants were enrolled from 04 December 2012 to 30 September 2014.
  The study consisted of a 24-week double-blind treatment period, a 108-week open-label treatment period, and a safety follow-up period.
Pre-assignment Details: Participants were to be randomly assigned in a 2:1:2:1 ratio to 1 of 4 treatment groups. Due to a misalignment error, some participants were erroneously assigned to incorrect treatment resulting in a final randomization ratio different from that originally stipulated in the protocol.
Groups:
- Placebo/Abrilumab 210 mg Q3M: Participants randomized to receive placebo by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks thereafter until week 24.
  During the open-label period, participants received abrilumab 210 mg once every 3 months (Q3M) for 108 weeks.
- Abrilumab 21 mg Q4W/Abrilumab 210 mg Q3M: Participants randomized to receive 21 mg abrilumab by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks (Q4W) thereafter until week 24.
  During the open-label period, participants received abrilumab 210 mg once every 3 months for 108 weeks.
- Abrilumab 70 mg Q4W/Abrilumab 210 mg Q3M: Participants randomized to receive 70 mg abrilumab by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks thereafter until week 24.
  During the open-label period, participants received abrilumab 210 mg once every 3 months for 108 weeks.
- Abrilumab 210 mg/Abrilumab 210 mg Q3M: Participants randomized to receive a single dose of 210 mg abrilumab by subcutaneous injection on day 1, followed by placebo at week 2, week 4, and every 4 weeks thereafter until week 24.
  During the open-label period, participants received abrilumab 210 mg once every 3 months for 108 weeks.
Period: Overall Study
Arm/Group | Placebo/Abrilumab 210 mg Q3M | Abrilumab 21 mg Q4W/Abrilumab 210 mg Q3M | Abrilumab 70 mg Q4W/Abrilumab 210 mg Q3M | Abrilumab 210 mg/Abrilumab 210 mg Q3M
Started | 100 | 27 | 85 | 42
Received Study Drug | 98 | 26 | 84 | 41
Entered Open-label Period | 84 | 21 | 75 | 37
Completed (Participants who completed the safety follow-up period) | 69 | 20 | 59 | 28
Not Completed | 31 | 7 | 26 | 14
Not completed — Withdrawal by Subject | 19 | 5 | 19 | 11
Not completed — Decision by Sponsor | 3 | 1 | 2 | 2
Not completed — Lost to Follow-up | 9 | 1 | 4 | 1
Not completed — Death | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants randomized to receive placebo by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks thereafter until week 24 during the double-blind treatment period.
- Abrilumab 21 mg Q4W: Participants randomized to receive 21 mg abrilumab by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks (Q4W) thereafter until week 24 during the double-blind treatment period.
- Abrilumab 70 mg Q4W: Participants randomized to receive 70 mg abrilumab by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks thereafter until week 24 during the double-blind treatment period.
- Abrilumab 210 mg: Participants randomized to receive a single dose of 210 mg abrilumab by subcutaneous injection on day 1, followed by placebo at week 2, week 4, and every 4 weeks thereafter until week 24 during the double-blind treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo | Abrilumab 21 mg Q4W | Abrilumab 70 mg Q4W | Abrilumab 210 mg | Total
Number analyzed (Participants) | 100 | 27 | 85 | 42 | 254
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (11.2) | 38.9 (14.2) | 35.6 (11.8) | 36.5 (9.4) | 36.4 (11.4)
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 99 | 27 | 85 | 42 | 253
  ≥ 65 years | 1 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 12 | 51 | 23 | 144
  Male | 42 | 15 | 34 | 19 | 110
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 100 | 26 | 85 | 41 | 252
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 1 | 1
  Black or African American | 2 | 0 | 0 | 1 | 3
  White | 97 | 26 | 82 | 40 | 245
  Other | 1 | 1 | 3 | 0 | 5
Any Prior Anti-Tumor Necrosis Factor (TNF) Use [Count of Participants; unit: Participants]
  Yes | 80 | 21 | 67 | 33 | 201
  No | 20 | 6 | 18 | 9 | 53
Enrollment Prior to Protocol Amendment 3 [Count of Participants; unit: Participants]
  Yes | 44 | 0 | 29 | 16 | 89
  No | 56 | 27 | 56 | 26 | 165
Duration of Crohn's Diease [Mean (Standard Deviation); unit: years] | 11.07 (8.33) | 12.58 (9.55) | 10.69 (7.75) | 11.31 (7.54) | 11.15 (8.12)
Crohn's Disease Activity Index (CDAI) Score [Mean (Standard Deviation); unit: units on a scale] — The CDAI is a weighted, composite index of 8 disease variables (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extra-intestinal manifestations or fistula, use or non-use of antidiarrheal agents, presence or absence of an abdominal mass, hematocrit, and body weight). Scores range from approximately 0 to 600, with a higher score indicating more-severe disease activity. Patients with scores of > 450 are considered to have very severe disease. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 99 | 27 | 84 | 42 | 252
    (all) | 303.8 (63.2) | 310.0 (83.5) | 314.0 (60.4) | 319.3 (67.5) | 310.5 (65.3)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Remission at Week 8
Description: Remission was defined as a Crohn's Disease Activity Index (CDAI) score < 150 at week 8.
  The CDAI is a weighted, composite index of 8 disease variables (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extra-intestinal manifestations or fistula, use or non-use of antidiarrheal agents, presence or absence of an abdominal mass, hematocrit, and body weight). Scores range from approximately 0 to 600, with a higher score indicating more-severe disease activity.
  The remission rate (percentage of participants with remission) was calculated based on observed data (unadjusted remission rate) and also after applying a logistic regression model including the factors of treatment group, stratification factors (prior anti-TNF use and pre- versus post-Protocol Amendment 3) and baseline CDAI Score (adjusted remission rate).
Time Frame: Week 8
Population: The full analysis set includes all randomized participants who received at least 1 dose of study drug. Both unadjusted and adjusted remission rates were calculated using non-responder imputation, where participants with a missing CDAI Score at week 8 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Abrilumab 21 mg Q4W | Abrilumab 70 mg Q4W | Abrilumab 210 mg
Number analyzed (Participants) | 98 | 26 | 84 | 41
percentage of participants
  Unadjusted remission rate | 13.3 | 23.1 | 14.3 | 19.5
  Adjusted remission rate | 12.8 | 23.1 | 14.4 | 21.9
Statistical Analysis 1: Comparison: Placebo vs Abrilumab 70 mg Q4W; Comparisons between treatment groups were made using remission rates estimated from a logistic regression model adjusted for baseline CDAI score and stratification factors (prior vs no prior TNF antagonist use and enrollment pre- vs post-protocol amendment); Test type: Superiority — The study was powered for formal statistical testing of the abrilumab 70 mg group. The primary and key secondary endpoints were tested under a sequential framework of statistical hypotheses, each with 2-sided significance level of 0.10 for the treatment effect of abrilumab 70 mg compared with placebo; p = 0.76, Regression, Logistic; Adjusted for baseline CDAI score and stratification factors; Odds Ratio (OR) = 1.15, 90% CI 2-sided [0.54 to 2.44] — An odds ratio > 1.0 indicates a higher remission rate for the abrilumab treatment group relative to placebo
Statistical Analysis 2: Comparison: Placebo vs Abrilumab 70 mg Q4W; The difference in remission rates, estimated from a logistic regression model adjusted for baseline CDAI score and stratification factors (prior vs no prior TNF antagonist use and enrollment pre- vs post-protocol amendment); Test type: Superiority; Difference in Adjusted Remission Rates = 1.6, 90% CI 2-sided [-7.9 to 8.9]
Statistical Analysis 3: Comparison: Placebo vs Abrilumab 210 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Analysis was not part of the formal testing; p = 0.22, Regression, Logistic; Adjusted for baseline CDAI score and stratification factors; Odds Ratio (OR) = 1.91, 90% CI 2-sided [0.80 to 4.57] — An odds ratio > 1.0 indicates a higher remission rate for the abrilumab treatment group relative to placebo
Statistical Analysis 4: Comparison: Placebo vs Abrilumab 210 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — Analysis was not part of the formal testing; Difference in Adjusted Remission Rates = 9.1, 90% CI 2-sided [-4.6 to 19.4]
Statistical Analysis 5: Comparison: Placebo vs Abrilumab 21 mg Q4W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Analysis was not part of the formal testing; p = 0.25, Regression, Logistic; Adjusted for baseline total CDAI score and stratification factors; Odds Ratio (OR) = 2.05, 90% CI 2-sided [0.74 to 5.73] — An odds ratio > 1.0 indicates a higher remission rate for the abrilumab treatment group relative to placebo
Statistical Analysis 6: Comparison: Placebo vs Abrilumab 21 mg Q4W; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — Analysis was not part of the formal testing; Difference in Adjusted Remission Rates = 10.3, 90% CI 2-sided [-6.8 to 22.6]

2. Secondary Outcome: Percentage of Participants With Remission at Week 12
Description: Remission was defined as a Crohn's Disease Activity Index (CDAI) score < 150. The CDAI is a weighted, composite index of 8 disease variables (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extra-intestinal manifestations or fistula, use or non-use of antidiarrheal agents, presence or absence of an abdominal mass, hematocrit, and body weight). Scores range from approximately 0 to 600, with a higher score indicating more-severe disease activity.
  The remission rate (percentage of participants with remission) was calculated based on observed data (unadjusted remission rate) and also after applying a logistic regression model including the factors of treatment group, stratification factors (prior anti-TNF use and pre- versus post-Protocol Amendment 3) and baseline CDAI Score (adjusted remission rate).
Time Frame: Week 12
Population: The full analysis set includes all randomized participants who received at least 1 dose of study drug. Both unadjusted and adjusted remission rates were calculated using non-responder imputation, where participants with a missing CDAI Score at week 12 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Abrilumab 21 mg Q4W | Abrilumab 70 mg Q4W | Abrilumab 210 mg
Number analyzed (Participants) | 98 | 26 | 84 | 41
percentage of participants
  Unadjusted remission rate | 18.1 | 33.3 | 25.3 | 27.0
  Adjusted remission rate | 20.1 | 43.8 | 31.0 | 34.8
Statistical Analysis 1: Comparison: Placebo vs Abrilumab 70 mg Q4W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.16, Regression, Logistic; Adjusted for baseline CDAI score and stratification factors; Odds Ratio (OR) = 1.78, 90% CI 2-sided [0.90 to 3.53] — An odds ratio > 1.0 indicates a higher remission rate for the abrilumab treatment group relative to placebo
Statistical Analysis 2: Comparison: Placebo vs Abrilumab 70 mg Q4W; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Difference in Adjusted Remission Rates = 10.9, 90% CI 2-sided [-1.8 to 21.0]
Statistical Analysis 3: Comparison: Placebo vs Abrilumab 210 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Analysis was not part of the formal testing; p = 0.13, Regression, Logistic; Adjusted for baseline CDAI score and stratification factors; Odds Ratio (OR) = 2.12, 90% CI 2-sided [0.93 to 4.84] — An odds ratio > 1.0 indicates a higher remission rate for the abrilumab treatment group relative to placebo
Statistical Analysis 4: Comparison: Placebo vs Abrilumab 210 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — Analysis was not part of the formal testing; Difference in Adjusted Remission Rates = 14.7, 90% CI 2-sided [-2.1 to 27.5]
Statistical Analysis 5: Comparison: Placebo vs Abrilumab 21 mg Q4W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Analysis was not part of the formal testing; p = 0.056, Regression, Logistic; Adjusted for baseline total CDAI score and stratification factors; Odds Ratio (OR) = 3.10, 90% CI 2-sided [1.17 to 8.20] — An odds ratio > 1.0 indicates a higher remission rate for the abrilumab treatment group relative to placebo
Statistical Analysis 6: Comparison: Placebo vs Abrilumab 21 mg Q4W; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — Analysis was not part of the formal testing; Difference in Adjusted Remission Rates = 23.7, 90% CI 2-sided [2.8 to 39.2]

3. Secondary Outcome: Percentage of Participants With Response at Week 12
Description: Response was defined as either remission (a CDAI score < 150) or a decrease from baseline in the CDAI score of ≥ 100 points.
  The CDAI is a weighted, composite index of 8 disease variables (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extra-intestinal manifestations or fistula, use or non-use of antidiarrheal agents, presence or absence of an abdominal mass, hematocrit, and body weight). Scores range from approximately 0 to 600, with a higher score indicating more-severe disease activity.
  The response rate (percentage of participants with response) was calculated based on observed data (unadjusted response rate) and also after applying a logistic regression model including the factors of treatment group, stratification factors (prior anti-TNF use and pre- versus post-Protocol Amendment 3) and baseline CDAI score (adjusted response rate).
Time Frame: Baseline and week 12
Population: The full analysis set includes all randomized participants who received at least 1 dose of study drug. Both unadjusted and adjusted response rates were calculated using non-responder imputation, where participants with a missing CDAI Score at week 12 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Abrilumab 21 mg Q4W | Abrilumab 70 mg Q4W | Abrilumab 210 mg
Number analyzed (Participants) | 98 | 26 | 84 | 41
percentage of participants
  Unadjusted response rate | 27.7 | 41.7 | 45.3 | 43.2
  Adjusted response rate | 35.3 | 50.4 | 55.1 | 50.9
Statistical Analysis 1: Comparison: Placebo vs Abrilumab 70 mg Q4W; Comparisons between treatment groups were made using response rates estimated from a logistic regression model adjusted for baseline CDAI score and stratification factors (prior vs no prior TNF antagonist use and enrollment pre- vs post-protocol amendment); Test type: Superiority; p = 0.021, Regression, Logistic; Adjusted for baseline CDAI score and stratification factors; Odds Ratio (OR) = 2.25, 90% CI 2-sided [1.27 to 4.01] — An odds ratio > 1.0 indicates a higher response rate for the abrilumab treatment group relative to placebo
Statistical Analysis 2: Comparison: Placebo vs Abrilumab 70 mg Q4W; The difference in response rates, estimated from a logistic regression model adjusted for baseline CDAI score and stratification factors (prior vs no prior TNF antagonist use and enrollment pre- vs post-protocol amendment); Test type: Superiority; Difference in Adjusted Response Rates = 19.8, 90% CI 2-sided [5.8 to 31.3]
Statistical Analysis 3: Comparison: Placebo vs Abrilumab 210 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — Analysis was not part of the formal testing; p = 0.14, Regression, Logistic; Adjusted for baseline CDAI score and stratification factors; Odds Ratio (OR) = 1.90, 90% CI 2-sided [0.94 to 3.87] — An odds ratio > 1.0 indicates a higher response rate for the abrilumab treatment group relative to placebo
Statistical Analysis 4: Comparison: Placebo vs Abrilumab 210 mg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority — Analysis was not part of the formal testing; Difference in Adjusted Response Rates = 15.7, 90% CI 2-sided [-2.3 to 29.7]
Statistical Analysis 5: Comparison: Placebo vs Abrilumab 21 mg Q4W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — Analysis was not part of the formal testing; p = 0.23, Regression, Logistic; Adjusted for baseline total CDAI score and stratification factors; Odds Ratio (OR) = 1.87, 90% CI 2-sided [0.79 to 4.39] — An odds ratio > 1.0 indicates a higher response rate for the abrilumab treatment group relative to placebo
Statistical Analysis 6: Comparison: Placebo vs Abrilumab 21 mg Q4W; [analysis description as in outcome 3, analysis 2]; Test type: Superiority — Analysis was not part of the formal testing; Difference in Adjusted Response Rates = 15.1, 90% CI 2-sided [-6.4 to 31.3]

4. Secondary Outcome: Percentage of Participants With Response at Week 8
Description: as for outcome 3
Time Frame: Baseline and week 8
Population: The full analysis set includes all randomized participants who received at least 1 dose of study drug. Both unadjusted and adjusted response rates were calculated using non-responder imputation, where participants with a missing CDAI Score at week 8 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Abrilumab 21 mg Q4W | Abrilumab 70 mg Q4W | Abrilumab 210 mg
Number analyzed (Participants) | 98 | 26 | 84 | 41
percentage of participants
  Unadjusted response rate | 26.4 | 33.3 | 42.9 | 30.6
  Adjusted response rate | 30.6 | 33.8 | 46.6 | 32.6
Statistical Analysis 1: Comparison: Placebo vs Abrilumab 70 mg Q4W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.047, Regression, Logistic; Adjusted for baseline CDAI score and stratification factors; Odds Ratio (OR) = 1.98, 90% CI 2-sided [1.13 to 3.47] — An odds ratio > 1.0 indicates a higher response rate for the abrilumab treatment group relative to placebo
Statistical Analysis 2: Comparison: Placebo vs Abrilumab 70 mg Q4W; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; Difference in Adjusted Response Rates = 16.0, 90% CI 2-sided [2.4 to 27.1]
Statistical Analysis 3: Comparison: Placebo vs Abrilumab 210 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — Analysis was not part of the formal testing; p = 0.84, Regression, Logistic; Adjusted for baseline CDAI score and stratification factors; Odds Ratio (OR) = 1.09, 90% CI 2-sided [0.52 to 2.29] — An odds ratio > 1.0 indicates a higher response rate for the abrilumab treatment group relative to placebo
Statistical Analysis 4: Comparison: Placebo vs Abrilumab 210 mg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority — Analysis was not part of the formal testing; Difference in Adjusted Response Rates = 1.9, 90% CI 2-sided [-15.2 to 15.2]
Statistical Analysis 5: Comparison: Placebo vs Abrilumab 21 mg Q4W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — Analysis was not part of the formal testing; p = 0.78, Regression, Logistic; Adjusted for baseline total CDAI score and stratification factors; Odds Ratio (OR) = 1.15, 90% CI 2-sided [0.49 to 2.72] — An odds ratio > 1.0 indicates a higher response rate for the abrilumab treatment group relative to placebo
Statistical Analysis 6: Comparison: Placebo vs Abrilumab 21 mg Q4W; [analysis description as in outcome 3, analysis 2]; Test type: Superiority — Analysis was not part of the formal testing; Difference in Adjusted Response Rates = 3.1, 90% CI 2-sided [-17.4 to 18.3]

5. Secondary Outcome: Percentage of Participants With Sustained Remission at Both Week 12 and Week 24
Description: Remission was defined as a Crohn's Disease Activity Index (CDAI) score < 150. Sustained remission was defined as achieving the criteria for remission at both week 12 and week 24.
  The CDAI is a weighted, composite index of 8 disease variables (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extra-intestinal manifestations or fistula, use or non-use of antidiarrheal agents, presence or absence of an abdominal mass, hematocrit, and body weight). Scores range from approximately 0 to 600, with a higher score indicating more-severe disease activity.
  The remission rate (percentage of participants with sustained remission) was calculated based on observed data (unadjusted remission rate) and also after applying a logistic regression model including the factors of treatment group, stratification factors (prior anti-TNF use and pre- versus post-Protocol Amendment 3) and baseline CDAI Score (adjusted remission rate).
Time Frame: Week 12 and week 24
Population: The full analysis set includes all randomized participants who received at least 1 dose of study drug. Both unadjusted and adjusted sustained remission rates were calculated using non-responder imputation, where participants with missing CDAI scores at week 12 or week 24 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Abrilumab 21 mg Q4W | Abrilumab 70 mg Q4W | Abrilumab 210 mg
Number analyzed (Participants) | 98 | 26 | 84 | 41
percentage of participants
  Unadjusted remission rate | 8.2 | 19.2 | 11.9 | 17.1
  Adjusted remission rate | 9.0 | 25.0 | 14.0 | 21.7
Statistical Analysis 1: Comparison: Placebo vs Abrilumab 70 mg Q4W; Comparisons between treatment groups were made using sustained remission rates estimated from a logistic regression model adjusted for baseline CDAI score and stratification factors (prior vs no prior TNF antagonist use and enrollment pre- vs post-protocol amendment); Test type: Superiority; p = 0.34, Regression, Logistic; Adjusted for baseline CDAI score and stratification factors; Odds Ratio (OR) = 1.65, 90% CI 2-sided [0.69 to 3.91] — An odds ratio > 1.0 indicates a higher sustained remission rate for the abrilumab treatment group relative to placebo
Statistical Analysis 2: Comparison: Placebo vs Abrilumab 70 mg Q4W; The difference in sustained remission rates, estimated from a logistic regression model adjusted for baseline CDAI score and stratification factors (prior vs no prior TNF antagonist use and enrollment pre- vs post-protocol amendment); Test type: Superiority; Difference in Adjusted Remission Rates = 5.0, 90% CI 2-sided [-3.9 to 11.7]
Statistical Analysis 3: Comparison: Placebo vs Abrilumab 210 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority — Analysis was not part of the formal testing; p = 0.078, Regression, Logistic; Adjusted for baseline CDAI score and stratification factors; Odds Ratio (OR) = 2.82, 90% CI 2-sided [1.07 to 7.41] — An odds ratio > 1.0 indicates a higher sustained remission rate for the abrilumab treatment group relative to placebo
Statistical Analysis 4: Comparison: Placebo vs Abrilumab 210 mg; [analysis description as in outcome 5, analysis 2]; Test type: Superiority — Analysis was not part of the formal testing; Difference in Adjusted Remission Rates = 12.8, 90% CI 2-sided [-0.6 to 22.6]
Statistical Analysis 5: Comparison: Placebo vs Abrilumab 21 mg Q4W; [analysis description as in outcome 5, analysis 1]; Test type: Superiority — Analysis was not part of the formal testing; p = 0.083, Regression, Logistic; Adjusted for baseline total CDAI score and stratification factors; Odds Ratio (OR) = 3.37, 90% CI 2-sided [1.07 to 10.66] — An odds ratio > 1.0 indicates a higher sustained remission rate for the abrilumab treatment group relative to placebo
Statistical Analysis 6: Comparison: Placebo vs Abrilumab 21 mg Q4W; [analysis description as in outcome 5, analysis 2]; Test type: Superiority — Analysis was not part of the formal testing; Difference in Adjusted Remission Rates = 16.0, 90% CI 2-sided [-1.2 to 28.3]

6. Secondary Outcome: Percentage of Participants With Sustained Remission at Both Week 8 and Week 24
Description: Remission was defined as a Crohn's Disease Activity Index (CDAI) score < 150. Sustained remission was defined as achieving the criteria for remission at both week 8 and week 24.
  The CDAI is a weighted, composite index of 8 disease variables (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extra-intestinal manifestations or fistula, use or non-use of antidiarrheal agents, presence or absence of an abdominal mass, hematocrit, and body weight). Scores range from approximately 0 to 600, with a higher score indicating more-severe disease activity.
  The remission rate (percentage of participants with sustained remission) was calculated based on observed data (unadjusted remission rate) and also after applying a logistic regression model including the factors of treatment group, stratification factors (prior anti-TNF use and pre- versus post-Protocol Amendment 3) and baseline CDAI Score (adjusted remission rate).
Time Frame: Week 8 and week 24
Population: The full analysis set includes all randomized participants who received at least 1 dose of study drug. Both unadjusted and adjusted sustained remission rates were calculated using non-responder imputation, where participants with missing CDAI scores at week 8 or week 24 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Abrilumab 21 mg Q4W | Abrilumab 70 mg Q4W | Abrilumab 210 mg
Number analyzed (Participants) | 98 | 26 | 84 | 41
percentage of participants
  Unadjusted remission rate | 7.1 | 15.4 | 9.5 | 12.2
  Adjusted remission rate | 5.9 | 14.3 | 8.7 | 12.7
Statistical Analysis 1: Comparison: Placebo vs Abrilumab 70 mg Q4W; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.47, Regression, Logistic; Adjusted for baseline CDAI score and stratification factors; Odds Ratio (OR) = 1.52, 90% CI 2-sided [0.59 to 3.93] — An odds ratio > 1.0 indicates a higher sustained remission rate for the abrilumab treatment group relative to placebo
Statistical Analysis 2: Comparison: Placebo vs Abrilumab 70 mg Q4W; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; Difference in Adjusted Remission Rates = 2.8, 90% CI 2-sided [-4.7 to 8.1]
Statistical Analysis 3: Comparison: Placebo vs Abrilumab 210 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority — Analysis was not part of the formal testing; p = 0.21, Regression, Logistic; Adjusted for baseline CDAI score and stratification factors; Odds Ratio (OR) = 2.32, 90% CI 2-sided [0.77 to 6.98] — An odds ratio > 1.0 indicates a higher sustained remission rate for the abrilumab treatment group relative to placebo
Statistical Analysis 4: Comparison: Placebo vs Abrilumab 210 mg; [analysis description as in outcome 5, analysis 2]; Test type: Superiority — Analysis was not part of the formal testing; Difference in Adjusted Remission Rates = 6.8, 90% CI 2-sided [-4.3 to 14.5]
Statistical Analysis 5: Comparison: Placebo vs Abrilumab 21 mg Q4W; [analysis description as in outcome 5, analysis 1]; Test type: Superiority — Analysis was not part of the formal testing; p = 0.21, Regression, Logistic; Adjusted for baseline total CDAI score and stratification factors; Odds Ratio (OR) = 2.66, 90% CI 2-sided [0.75 to 9.45] — An odds ratio > 1.0 indicates a higher sustained remission rate for the abrilumab treatment group relative to placebo
Statistical Analysis 6: Comparison: Placebo vs Abrilumab 21 mg Q4W; [analysis description as in outcome 5, analysis 2]; Test type: Superiority — Analysis was not part of the formal testing; Difference in Adjusted Remission Rates = 8.4, 90% CI 2-sided [-6.0 to 17.9]

7. Secondary Outcome: Change From Baseline in CDAI Score at Week 12
Description: The CDAI is a weighted, composite index of 8 disease variables (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extra-intestinal manifestations or fistula, use or non-use of antidiarrheal agents, presence or absence of an abdominal mass, hematocrit, and body weight). Scores range from approximately 0 to 600, with a higher score indicating more-severe disease activity.
Time Frame: Baseline and week 12
Population: The full analysis set includes all randomized participants who received at least 1 dose of study drug. Missing data were handled using the inverse probability weighting (IPW) method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Abrilumab 21 mg Q4W | Abrilumab 70 mg Q4W | Abrilumab 210 mg
Number analyzed (Participants) | 98 | 26 | 84 | 41
units on a scale | -55.32 (11.41) | -92.16 (21.85) | -97.41 (12.92) | -96.11 (22.78)
Statistical Analysis 1: Comparison: Placebo vs Abrilumab 70 mg Q4W; Comparisons between treatment arms was conducted using an inverse probability weighting (IPW) generalized estimating equations (GEE) model adjusted for prior anti-TNF use, pre-versus post-protocol amendment 3 and baseline CDAI score; Test type: Superiority; p = 0.006, IPW GEE Model; Adjusted for prior anti-TNF use, pre-versus post-protocol amendment 3 and baseline CDAI score; LS Mean Treatment Difference = -42.09, 90% CI 2-sided [-67.3 to -16.9]
Statistical Analysis 2: Comparison: Placebo vs Abrilumab 210 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority — Analysis was not part of the formal testing; p = 0.095, IPW GEE Model; Adjusted for prior anti-TNF use, pre-versus post-protocol amendment 3 and baseline CDAI score; LS Mean Treatment Difference = -40.79, 90% CI 2-sided [-81.5 to -0.5]
Statistical Analysis 3: Comparison: Placebo vs Abrilumab 21 mg Q4W; [analysis description as in outcome 7, analysis 1]; Test type: Superiority — Analysis was not part of the formal testing; p = 0.11, IPW GEE Model; Adjusted for prior anti-TNF use, pre-versus post-protocol amendment 3 and baseline CDAI score; LS Mean Treatment Difference = -36.84, 90% CI 2-sided [-74.3 to 0.7]

8. Secondary Outcome: Change From Baseline in CDAI Score at Week 8
Description: as for outcome 7
Time Frame: Baseline and week 8
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Abrilumab 21 mg Q4W | Abrilumab 70 mg Q4W | Abrilumab 210 mg
Number analyzed (Participants) | 98 | 26 | 84 | 41
units on a scale | -64.05 (9.62) | -80.42 (20.86) | -91.52 (11.78) | -87.64 (19.89)
Statistical Analysis 1: Comparison: Placebo vs Abrilumab 70 mg Q4W; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.045, IPW GEE Model; Adjusted for prior anti-TNF use, pre-versus post-protocol amendment 3 and baseline CDAI score; LS Mean Treatment Difference = -27.47, 90% CI 2-sided [-50.0 to -4.9]
Statistical Analysis 2: Comparison: Placebo vs Abrilumab 210 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority — Analysis was not part of the formal testing; p = 0.27, IPW GEE Model; Adjusted for prior anti-TNF use, pre-versus post-protocol amendment 3 and baseline CDAI score; LS Mean Treatment Difference = -23.59, 90% CI 2-sided [-58.7 to 11.5]
Statistical Analysis 3: Comparison: Placebo vs Abrilumab 21 mg Q4W; [analysis description as in outcome 7, analysis 1]; Test type: Superiority — Analysis was not part of the formal testing; p = 0.45, IPW GEE Model; Adjusted for prior anti-TNF use, pre-versus post-protocol amendment 3 and baseline CDAI score; LS Mean Treatment Difference = -16.37, 90% CI 2-sided [-51.8 to 19.1]

ADVERSE EVENTS:
Time Frame: From first dose of study drug to week 24 in the double-blind period and from first dose of study drug in the open-label period to 12 weeks after last dose in the open-label period (up to 108 weeks).
Description: One participant randomized to the 21 mg abrilumab treatment group received 70 mg abrilumab in error and is counted in the Abrilumab 70 mg group for safety analyses in both treatment periods.
  Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- DB Period: Placebo: Participants received placebo by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks thereafter until week 24 during the double-blind (DB) treatment period.
- DB Period: Abrilumab 21 mg Q4W: Participants received 21 mg abrilumab by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks thereafter until week 24 during the double-blind treatment period.
- DB Period: Abrilumab 70 mg Q4W: Participants received 70 mg abrilumab by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks thereafter until week 24 during the double-blind treatment period.
- DB Period: Abrilumab 210 mg: Participants received a single dose of 210 mg abrilumab by subcutaneous injection on day 1, followed by placebo at week 2, week 4, and every 4 weeks thereafter until week 24 during the double-blind treatment period.
- OL Period: Placebo/Abrilumab 210 mg Q3M: Participants who received placebo during the double-blind treatment period received abrilumab 210 mg once every 3 months (Q3M) for 108 weeks during the open-label (OL) treatment period.
- OL Period: Abrilumab 21 mg Q4W/210 mg Q3M: During the open-label period, participants who received 21 mg abrilumab Q4W during the DB treatment period received abrilumab 210 mg once every 3 months for 108 weeks.
- OL Period: Abrilumab 70 mg Q4W/210 mg Q3M: Participants who received 70 mg abrilumab Q4W during the DB treatment period received abrilumab 210 mg once every 3 months for 108 weeks during the open-label period.
- Period: Abrilumab 210 mg/210 mg Q3M: Participants who received 210 mg abrilumab during the DB treatment period received abrilumab 210 mg once every 3 months for 108 weeks during the open-label period.
Arm/Group | DB Period: Placebo | DB Period: Abrilumab 21 mg Q4W | DB Period: Abrilumab 70 mg Q4W | DB Period: Abrilumab 210 mg | OL Period: Placebo/Abrilumab 210 mg Q3M | OL Period: Abrilumab 21 mg Q4W/210 mg Q3M | OL Period: Abrilumab 70 mg Q4W/210 mg Q3M | Period: Abrilumab 210 mg/210 mg Q3M
Serious Adverse Events (participants affected / at risk) | 14/98 | 7/25 | 13/85 | 6/41 | 24/84 | 3/20 | 19/76 | 12/37
Other Adverse Events (participants affected / at risk) | 61/98 | 14/25 | 48/85 | 27/41 | 61/84 | 16/20 | 55/76 | 28/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB Period: Placebo (N=98) | DB Period: Abrilumab 21 mg Q4W (N=25) | DB Period: Abrilumab 70 mg Q4W (N=85) | DB Period: Abrilumab 210 mg (N=41) | OL Period: Placebo/Abrilumab 210 mg Q3M (N=84) | OL Period: Abrilumab 21 mg Q4W/210 mg Q3M (N=20) | OL Period: Abrilumab 70 mg Q4W/210 mg Q3M (N=76) | Period: Abrilumab 210 mg/210 mg Q3M (N=37)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 9 | 4 | 3 | 2 | 9 | 2 | 8 | 6
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Enterocolonic fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ileal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 3 | 1 | 0 | 0 | 1 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Abdominal wall abscess (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abscess intestinal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
External ear cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intrauterine infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Perineal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia parainfluenzae viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Psoas abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Retroperitoneal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tubo-ovarian abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulval abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aborted pregnancy (Social circumstances) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Ileocolectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Scoliosis surgery (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB Period: Placebo (N=98) | DB Period: Abrilumab 21 mg Q4W (N=25) | DB Period: Abrilumab 70 mg Q4W (N=85) | DB Period: Abrilumab 210 mg (N=41) | OL Period: Placebo/Abrilumab 210 mg Q3M (N=84) | OL Period: Abrilumab 21 mg Q4W/210 mg Q3M (N=20) | OL Period: Abrilumab 70 mg Q4W/210 mg Q3M (N=76) | Period: Abrilumab 210 mg/210 mg Q3M (N=37)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 3 | 2 | 3 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 3 | 0 | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 9 | 1 | 8 | 1 | 9 | 2 | 10 | 2
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 3 | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 2 | 1 | 1 | 2 | 2 | 1 | 2 | 1
Crohn's disease (Gastrointestinal disorders) | 8 | 1 | 2 | 2 | 14 | 1 | 12 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 4 | 2 | 5 | 0 | 5 | 2
Gastrointestinal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 1 | 2 | 3 | 7 | 2 | 5 | 4
Oral discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 2
Vomiting (Gastrointestinal disorders) | 3 | 0 | 3 | 3 | 5 | 2 | 2 | 2
Asthenia (General disorders) | 2 | 1 | 1 | 1 | 5 | 0 | 1 | 2
Fatigue (General disorders) | 4 | 1 | 2 | 3 | 3 | 0 | 1 | 0
Influenza like illness (General disorders) | 4 | 3 | 4 | 0 | 5 | 1 | 7 | 3
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1 | 3 | 1 | 1 | 0 | 1
Pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 2 | 4 | 2 | 4 | 3 | 2 | 5
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 1 | 2 | 0 | 1 | 0 | 4 | 0
Bronchitis (Infections and infestations) | 2 | 1 | 3 | 2 | 4 | 1 | 2 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 1
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 6 | 0 | 3 | 1 | 2 | 0 | 7 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 1 | 3 | 4 | 1 | 10 | 6
Nasopharyngitis (Infections and infestations) | 11 | 2 | 7 | 3 | 12 | 2 | 14 | 6
Psoas abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 2 | 1 | 2 | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 7 | 1 | 6 | 0 | 2 | 3
Urinary tract infection (Infections and infestations) | 2 | 0 | 6 | 1 | 3 | 2 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 2 | 2 | 2 | 1 | 3 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood iron decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Clostridium test positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Magnesium deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1
Zinc deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 1 | 8 | 3 | 5 | 2 | 7 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 2 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 0 | 1 | 1 | 3 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 2 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 3 | 2 | 2 | 2 | 2
Dizziness (Nervous system disorders) | 7 | 1 | 4 | 2 | 0 | 0 | 2 | 1
Headache (Nervous system disorders) | 11 | 4 | 12 | 8 | 7 | 3 | 2 | 3
Memory impairment (Nervous system disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 2 | 2 | 7 | 2 | 4 | 0 | 1 | 2
Depression (Psychiatric disorders) | 2 | 0 | 0 | 1 | 1 | 2 | 2 | 3
Insomnia (Psychiatric disorders) | 3 | 1 | 1 | 0 | 3 | 0 | 5 | 2
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 4 | 2 | 4 | 1 | 1 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 1 | 1 | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 2 | 1 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1 | 6 | 0 | 2 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Female sterilisation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.